CLINICAL TRIAL: NCT05320731
Title: A Comparative Study Between Atomization and Nebulization for Airway Topicalization During Awake Nasotracheal Fiberoptic Intubation
Brief Title: Atomization Vs. Nebulization for Airway Topicalization During Awake Nasotracheal Fiberoptic Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ashraf Torki, Lecturer of Anesthesia, Zagazig University (Principal Investigator), Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZU-IRB #9351
Record Dates: First submitted 2022-03-23; First posted 2022-04-11 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Awake Fiberoptic Intubation
Keywords: Awake fiberoptic intubation; Nebulization; Atomization
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Both the anesthesiologist performing the fibroscopy and the data collector will be blind to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nebulization with lidocaine (Active Comparator): A face mask nebulizer with oxygen flow rate of 8 L/min will be used to deliver 10 mL of 2% lidocaine. Patients will be encouraged to inhale deeply to facilitate entrainment of nebulized LA into their airway. Adequate topical anesthesia will be confirmed by heaviness or numbness of the tongue.
  Interventions: Procedure: Nebulization with lidocaine
- Atomization with lidocaine (Active Comparator): Our simple atomization device, a modification of the McKenzie technique, will be used. One end of oxygen bubble tubing will be cut to fit into the barrel of 1 mL syringe and attached to one connector of a 3-way tap. A 10-mL syringe filled with 2% lidocaine will be attached to the other connector of the 3-way tap. A 6 Fr suction catheter, with its colored end cut and its distal blind end cut open, will be attached to oxygen bubble tubing via the male Luer connector of the 3-way tap. The other end of bubble tubing will be then attached to an oxygen source turned on to deliver a flow of 6 L/min. As LA is slowly atomized as a jet-like spray, the catheter will be directed towards the soft palate and posterior pharynx in a controlled fashion during patients' inspiration to topicalize the airway. Patients will be asked to take full vital capacity breaths of atomized LA contained oxygen. Adequate topical anesthesia will be confirmed by tongue heaviness or numbness
  Interventions: Procedure: Atomization with lidocaine

INTERVENTIONS:
Procedure: Nebulization with lidocaine — A face mask nebulizer with oxygen flow rate of 8 L/min will be used to deliver 10 mL of 2% lidocaine. Patients will be encouraged to inhale deeply to facilitate entrainment of nebulized LA into their airway. Adequate topical anesthesia will be confirmed by heaviness or numbness of the tongue.
  Arms: Nebulization with lidocaine
Procedure: Atomization with lidocaine — A simple atomization device as a modification of the McKenzie technique will be used. One end of oxygen bubble tubing will be cut to fit into the barrel of 1 mL syringe and attached to one connector of a 3-way tap. A 10-mL syringe filled with 2% lidocaine will be attached to the other connector of the 3-way tap. A 6 Fr suction catheter, with its colored end cut and its distal blind end cut open, will be attached to oxygen bubble tubing via the male Luer connector of the 3-way tap. The other end of bubble tubing will be then attached to an oxygen source turned on to deliver a flow of 6 L/min. As LA is slowly atomized as a jet-like spray, the catheter will be directed towards the soft palate and posterior pharynx in a controlled fashion during patients' inspiration to topicalize the airway. Patients will be asked to take full vital capacity breaths of atomized LA contained oxygen. Adequate topical anesthesia will be confirmed by tongue heaviness or numbness
  Arms: Atomization with lidocaine

SUMMARY:
Intubation of difficult airway is a challenge for anesthetist. There many causes of difficult airway, and previous studies concluded that awake fiber-optic intubation (AFOI) is the gold standard for the management of these patients. Several studies showed that airway nerve blocks provide rapid and deep airway anesthesia, however, due to their several disadvantages, topicalization of the airway represents a promising alternative to them. Some studies revealed that nebulization and atomization of the airway provide adequate anesthesia for AFOI. In the present study, we try to find out which is more effective for topicalization of the airway during nasotracheal AFOI; nebulization or atomization. We used a simple atomization device as a modification of the McKenzie technique.

DETAILED DESCRIPTION:
Site of the Study: Zagazig university surgical hospitals.

Type of the Study: Prospective randomized double-blinded clinical trial.

Withdrawal Criteria:

The patient has the right to withdraw from the study at any time without any negative consequences on medical or surgical treatment plan.

Randomization:

Group I: will receive Nebulization with lidocaine, Group II: will receive Atomization with lidocaine.

Computer-generated randomization numbers will be used to randomly assign patients into 2 groups using sealed opaque envelopes that will be randomly selected by each patient and contained a group number in which patient was enrolled. Once enrolled in the study, patients will be randomly assigned into 2 groups; Both the anesthesiologist performing the fibroscopy and the data collector will be blind to group assignment.

Type of the Study: Prospective randomized double-blinded clinical trial.

Steps of Performance:

Preoperative Assessment:

A thorough airway evaluation will be performed using the Simplified Airway Risk Index "SARI". Airway assessment also will include other causes of anticipated difficult intubation e.g., airway pathology, craniofacial abnormalities, or cervical spine instability.

All patients will be assessed by history taking, clinical examination and laboratory investigations, which will include; Complete blood count (CBC), Prothrombin time and concentration (PT and PC), Partial thromboplastin time (PTT), International normalized ratio (INR), liver and kidney function tests. Other investigations (e.g., electrocardiography, echocardiography, and chest x-ray) will be done according to patient's medical condition.

Preoperative Preparation:

Procedure explanation will be done the day before surgery, and informed written consent will be obtained from patients after discussing with them the cause of performing the procedure, its benefits and possible complications that may occur. Standard fasting guidelines will be also explained to the patients to be followed.

In the Procedure Area:

Premedication, nasal preparation and topicalization technique will be performed by independent anesthesiologist in the procedure area, where patient's vital signs are monitored, then the patient will be shifted to the operating room where fibroscopy and intubation will be performed by another blinded anesthesiologist. The procedure area will be equipped for emergency management and close monitoring of the patient.

A. Monitoring:

Monitoring will be applied and maintained throughout the procedure, including 5- lead electrocardiogram (ECG), non-invasive arterial blood pressure and pulse oximeter. Hemodynamic parameters heart rate (HR), mean arterial blood pressure (MAP), and oxygen saturation (SpO2) will be recorded, as baseline recordings before sedation and after Ramsay sedation score 2.

B. Premedication:

After ensuring of working 18 gauge intravenous (IV) line, All patients will receive IV bolus doses of the following; Atropine; as anti-sialogouge (0.5 mg IV). Midazolam; as sedative, starting dose from 20 up to 50 μg/kg. Fentanyl; as analgesic and antitussive, starting dose from 0.5 up to 1.5-µg/kg Midazolam and fentanyl doses will be titrated according to the patient's level of sedation with target to obtain a cooperative, oriented and tranquil patient (Ramsay sedation score of 2).

C. Nasal Preparation:

All patients' nostrils will be instilled with Xylometazoline 1% nasal drops (2-3 drop for each nostril). Anesthesia of the nasal mucosa will be achieved by application of 3 cotton swabs soaked in 2 mL of 2% lidocaine solution. The cotton swabs will be introduced into the preferred nostril, one at a depth of 1.5 cm superiorly (to block the branches of ethmoidal nerves), and two at a depth of 2-2.5 cm (to block the sphenopalatine ganglion and branches of the maxillary division of the trigeminal nerve). The swabs will be kept in place for 3 min.

The preferred nostril for FOI will be then progressively dilated with silicone nasopharyngeal airway starting 6.5 up to 7.5 mm smeared with 2% lidocaine jelly. The nasopharyngeal airway will be removed immediately before fibroscopy. This method allows for lubrication of the nasal passages and also ensures that these passages are patent and likely large enough for the ETT.

D. Topicalization Technique:

After ensuring adequate nasal preparation, the patient's envelope which contains the number of group will be opened and it will be recorded in the data collection sheet as a number of group because the data collector will be blind to the intervention which will be done to the patient, only the anesthetist knows each number will be referring to which intervention.

Group I: will receive Nebulization with lidocaine. Group II: will receive Atomization with lidocaine. To ensure investigator blinding, nebulization and atomization will be administered by an independent anesthesiologist, and the patient will be then moved from the procedure area to the operating room where, after recording the vital signs, another blinded senior anesthesiologist, with previous experience in FOI, will perform the procedure.

1. Nebulization Technique:

   A face mask nebulizer with oxygen flow rate of 8 L/min will be used to deliver 10 mL of 2% lidocaine. Patients will be encouraged to inhale deeply to facilitate entrainment of nebulized LA into their airway. Adequate topical anesthesia will be confirmed by heaviness or numbness of the tongue.
2. Atomization Technique:

Our simple atomization device, a modification of the McKenzie technique, will be used for atomization. One end of oxygen bubble tubing will be cut to fit into the barrel of 1 mL syringe which will be attached to one female Luer connector of a three-way tap. A 10-mL syringe filled with 2% lidocaine will be attached to the other female Luer connector of the three-way tap. A 6 French suction catheter, with its colored end cut and its distal blind end cut open, will be attached to oxygen bubble tubing via the male Luer connector of the three-way tap. The other end of bubble tubing will be then attached to an oxygen source, which will be turned on to deliver a flow of 6 L/min. As LA is slowly atomized as a jet-like spray, the suction catheter will be directed towards the soft palate and posterior pharynx in a controlled fashion during patients' inspiration to topicalize the airway. Patients will be asked to take full vital capacity breaths of atomized LA contained oxygen to anaesthetize pharynx, glottis and subglottic structures. The patient will be asked to gargle the lidocaine in the mouth for as long as possible. Adequate topical anesthesia will be confirmed by tongue heaviness or numbness.

In the Operating Room:

A. Monitoring:

The same monitoring as in the procedure area will be applied and maintained throughout the procedure, including 5- lead electrocardiogram (ECG), non-invasive arterial blood pressure, pulse oximeter, and capnography.

B. Fibroscopy & Intubation:

After ensuring adequate sedation and optimal topical anesthesia, a fiberoptic scope (Pentax® FI-16BS, 5.2mm; Japan) loaded with an appropriate size ETT (size 7.0-7.5 mm internal diameter for male patients and size 6.5-7.0 mm for female patients) will be inserted nasally into the chosen nostril after removal of the nasopharyngeal airway.

Supplemental oxygen (2 L/min) will be delivered through the working channel of the FOB for oxygenation and prevention of mucosal webbing of the tip of the instrument. Any hypoxic episode (SPO2 < 90%) during intubation will be recorded.

Supplemental LA will be given as 2 ml aliquots of 2% lidocaine through the working channel of FOB by spray-as-you-go technique (next aliquot given only after waiting for 30-60 sec.).

Bronchoscopy-guided intubation time will be calculated as the time from passing the flexible fiberoptic bronchoscope tip through the nostril to the first reading obtained by the capnograph after endotracheal intubation.

Once the position of the fiberscope in the trachea is confirmed, the tracheal tube will be railroaded and positioned approximately 3 cm above the carina and secured. After the confirmation of ETT position by auscultation and capnography, GA will be administered with Propofol 2 mg/ kg and Rocuronium 0.6 mg/kg IV were administered and the patient will be connected to the ventilator.

Total LA Dose:

The total dose of lidocaine administered will be limited to 6 mg/kg which is lesser than the maximum recommended dose.

Assessment of the Quality of AFOI:

The quality of AFOI will be measured using intubating condition score, vocal cord position score, intraoperative patient comfort score and postoperative patient satisfaction score, as shown below.

Intubating Condition Score:

1. Optimal; No hold-up or collision of tracheal tube with vocal cords.
2. Suboptimal; Hold-up relieved by one rotation of the tube.
3. Difficult; Hold-up requiring more than one rotation of the tube.
4. Failure; Failed attempt at awake fiberoptic intubation.

Vocal Cord Position Score:

1; Relaxed, 2; Partially Relaxed and 3; Adducted.

Intraoperative Patient Comfort Score:

A. Cough & Gag Severity:

1; None, 2; Minimal coughing or gagging (< 3 times) like "clearing throat", 3; Mild coughing or gagging lasting < 1 min., and 4; Persistent coughing or gagging.

B. Comfort during Intubation:

1; No reaction, 2; Slight grimacing, 3; Severe grimacing, 4; Verbal objection, and 5; Defensive movements of head, hands, or feet.

C. Post-intubation Assessment:

1; Cooperative, 2; Restless/minimal resistance, and 3; Severe resistance/ requirement for immediate general anesthesia.

Postoperative Patient Satisfaction Score:

1; Excellent, 2; Good, 3; Fair and 4: Poor.

Parameters including intubating condition and vocal cord position will be recorded by the anesthesiologist performing the fiberoptic bronchoscopy-guided intubation, while intubation time, patient comfort and vital signs will be recorded by another independent observer who will be blinded to group assignment.

Measured Parameters:

A. Hemodynamics; Hemodynamic parameters including; HR, MAP, and SpO2 will be recorded, at the following times:

1. Baseline recordings before sedation (T0).
2. After Ramsay sedation score 2 (T1).
3. At the beginning of the fibrescopy (T2).
4. After entry of the FOB in the trachea (T3).
5. After advancing the ETT through the nasopharynx (T4).
6. Immediately post-intubation (T5).
7. 1, 3 and 5 min. post-intubation (T6). Hemodynamic monitoring will be concluded 5 min. post intubation.

B. Bronchoscopy-guided Intubation Time; will be measured as the time from passing the flexible fiberoptic bronchoscope tip through the nostril to the first reading obtained by the capnograph after endotracheal intubation.

C. Quality of AFOI; will be measured by intubating condition score, vocal cord position score, intraoperative patient comfort score and postoperative patient satisfaction score.

D. Success Rate; Defined as successful intubation with confirmation of ETT position by capnography and auscultation and securing the ETT as the endpoint of the trial, otherwise, the case will be considered failed and will be excluded from the study.

Complications:

Hoarseness, sore throat or any signs of lidocaine toxicity such as tinnitus, perioral tingling, seizures or cardiovascular collapse, will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Consent obtained from all patients included in this study.
2. Age 18 - 60 years, of both sexes.
3. ASA class I, II and III.
4. Anticipated difficult airway; SARI score ≥ 4, airway pathology, craniofacial abnormalities, or cervical spine instability.
5. Scheduled for elective non-cardiac surgery requiring general anesthesia and endotracheal intubation.

Exclusion Criteria:

1. Patient refusal, uncooperative and mentally retarded patients.
2. Full stomach patients.
3. Patients with nasal fractures or trauma, fracture base of the skull, bleeding disorder, epistaxis or active oral bleeding.
4. Active cough or respiratory tract infection and bronchial asthma.
5. Allergy to lidocaine.
6. Raised intracranial pressure or intraocular pressure.
7. Cerebral aneurysm, history of recent acute myocardial infarction or cerebrovascular accident.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Bronchoscopy-guided intubation time | Intraoperative (during intubation)
  Time from passing the flexible fiberoptic bronchoscope tip through the nostril to the first reading obtained by the capnograph after endotracheal intubation

SECONDARY OUTCOMES:
Intubating Condition Score: | Intraoperative (during intubation)
  Optimal (Best); No hold-up or collision of tracheal tube with vocal cords. Suboptimal; Hold-up relieved by one rotation of the tube. Difficult; Hold-up requiring more than one rotation of the tube. Failure (Worst); Failed attempt at awake fiberoptic intubation.
Vocal Cord Position Score: | Intraoperative (during intubation)
  1; Relaxed (Best), 2; Partially Relaxed and 3; Adducted (Worst)
Intraoperative Patient Comfort Score: | Intraoperative (during and immediately post-intubation)
  A. Cough & Gag Severity:
  1; None (Best), 2; Minimal coughing or gagging (< 3 times) like "clearing throat", 3; Mild coughing or gagging lasting < 1 min., and 4; Persistent coughing or gagging (Worst).
  B. Comfort during Intubation:
  1; No reaction (Best), 2; Slight grimacing, 3; Severe grimacing, 4; Verbal objection, and 5; Defensive movements of headBest), hands, or feet (Worst).
  C. Post-intubation Assessment:
  1; Cooperative (Best), 2; Restless/minimal resistance, and 3; Severe resistance/ requirement for immediate general anesthesia (Worst).
Postoperative Patient Satisfaction Score: | Postoperative 24 hours
  1; Excellent (Best), 2; Good, 3; Fair and 4: Poor (Worst).

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf A Torki, MD, Principal Investigator — Anesthesia and surgical intensive care, zagazig university, faculty of medicine; Mona A Shahin, MD, Study Director — Anesthesia and surgical intensive care, zagazig university, faculty of medicine
Locations (1):
- Zagazig university hospitals, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ikeda S, Yanai N, Ishikawa S. Flexible bronchofiberscope. Keio J Med. 1968 Mar;17(1):1-16. doi: 10.2302/kjm.17.1. No abstract available. PMID 5674435
- [Background] Murphy P. A fibre-optic endoscope used for nasal intubation. Anaesthesia. 1967 Jul;22(3):489-91. doi: 10.1111/j.1365-2044.1967.tb02771.x. No abstract available. PMID 4951601
- [Background] Gupta B, Kohli S, Farooque K, Jalwal G, Gupta D, Sinha S, Chandralekha. Topical airway anesthesia for awake fiberoptic intubation: Comparison between airway nerve blocks and nebulized lignocaine by ultrasonic nebulizer. Saudi J Anaesth. 2014 Nov;8(Suppl 1):S15-9. doi: 10.4103/1658-354X.144056. PMID 25538514
- [Background] Dhasmana SC. Nasotracheal fiberoptic intubation: patient comfort, intubating conditions and hemodynamic stability during conscious sedation with different doses of dexmedetomidine. J Maxillofac Oral Surg. 2014 Mar;13(1):53-8. doi: 10.1007/s12663-012-0469-0. Epub 2013 Jan 18. PMID 24644397
- [Background] Kundra P, Kutralam S, Ravishankar M. Local anaesthesia for awake fibreoptic nasotracheal intubation. Acta Anaesthesiol Scand. 2000 May;44(5):511-6. doi: 10.1034/j.1399-6576.2000.00503.x. PMID 10786733
- [Background] Mathur PR, Jain N, Kumar A, Thada B, Mathur V, Garg D. Comparison between lignocaine nebulization and airway nerve block for awake fiberoptic bronchoscopy-guided nasotracheal intubation: a single-blind randomized prospective study. Korean J Anesthesiol. 2018 Apr;71(2):120-126. doi: 10.4097/kjae.2018.71.2.120. Epub 2018 Apr 2. PMID 29619784
- [Background] Techanivate A, Leelanukrom R, Prapongsena P, Terachinda D. Effectiveness of mouthpiece nebulization and nasal swab stick packing for topical anesthesia in awake fiberoptic nasotracheal intubation. J Med Assoc Thai. 2007 Oct;90(10):2063-71. PMID 18041425
- [Background] Mostafa SM, Murthy BV, Hodgson CA, Beese E. Nebulized 10% lignocaine for awake fibreoptic intubation. Anaesth Intensive Care. 1998 Apr;26(2):222-3. No abstract available. PMID 9564411
- [Background] Ahmed I. Regional and Topical Anesthesia for Awake Endotracheal Intubation. In: Hadzic's Textbook of Regional Anesthesia and Acute Pain Management, 2nd ed: McGraw Hill Professional. 2017:20;289-99.
- [Background] Sinha S, Chakraborty, Mondal A, et al. (2019). Comparative study of nebulisation, airway nerve block and atomisation with lignocaine in topical airway anaesthesia for awake fibre-optic intubation. Journal of Evidence Based Medicine and Healthcare. 6. 1882-1886. 10.18410/jebmh/2019/383.
- [Background] Gjonaj ST, Lowenthal DB, Dozor AJ. Nebulized lidocaine administered to infants and children undergoing flexible bronchoscopy. Chest. 1997 Dec;112(6):1665-9. doi: 10.1378/chest.112.6.1665. PMID 9404766
- [Background] British Thoracic Society Bronchoscopy Guidelines Committee, a Subcommittee of Standards of Care Committee of British Thoracic Society. British Thoracic Society guidelines on diagnostic flexible bronchoscopy. Thorax. 2001 Mar;56 Suppl 1(Suppl 1):i1-21. doi: 10.1136/thorax.56.suppl_1.i1. No abstract available. PMID 11158709
- [Background] Reed AP. Preparation of the patient for awake flexible fiberoptic bronchoscopy. Chest. 1992 Jan;101(1):244-53. doi: 10.1378/chest.101.1.244. No abstract available. PMID 1729077
- [Background] Chavan G, Chavan AU, Patel S, Anjankar V, Gaikwad P. Airway Blocks Vs LA Nebulization- An interventional trial for Awake Fiberoptic Bronchoscope assisted Nasotracheal Intubation in Oral Malignancies. Asian Pac J Cancer Prev. 2020 Dec 1;21(12):3613-3617. doi: 10.31557/APJCP.2020.21.12.3613. PMID 33369459
- [Background] Yadav U, Kumar A, Gupta P. A Comparative Study of Airway Nerve Blocks and Atomized Lidocaine by the Laryngo-Tracheal Mucosal Atomization Device (LMA MADgic) Airway for Oral Awake Fiberoptic Intubation. Cureus. 2021 Jun 20;13(6):e15772. doi: 10.7759/cureus.15772. eCollection 2021 Jun. PMID 34295582